CLINICAL TRIAL: NCT04393961
Title: At-Home COVID-19 Antibody Test Usability Assessment & Behavior Change Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ProofPilot (Industry)
Collaborators: Radish Health (Unknown); Sanesco (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2458
Record Dates: First submitted 2020-04-24; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-04

CONDITIONS: COVID19; COVID-19; Coronavirus
Keywords: antibody; testing; remote trial
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This study will include four arms. The experiences across all 4 arms will be exactly the same. Each arm has a slightly different experience with COVID-19.
Masking Description: This is a device feasibility trial. There is no blinding or masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Past Positive COVID-19 confirmed (Other): Invited participants who Radish Health has completed a positive COVID-19 test who have recovered from all symptoms for more than 14 days.
  Interventions: Device: Premier Biotech COVID-19 IgG/IgM Rapid test Cassette
- Physician Diagnosed: Not Tested (Other): Individuals who self report that a medical professional has told them they likely have COVID-19 (and have since recovered), but did not get a confirmatory test.
  Interventions: Device: Premier Biotech COVID-19 IgG/IgM Rapid test Cassette
- Self-Diagnosed Not Tested (Other): Participant suspects they contracted (and have since recovered) from COVID-19, but they do not have a medical diagnosis or confirmatory test.
  Interventions: Device: Premier Biotech COVID-19 IgG/IgM Rapid test Cassette
- Likely Exposed, No Symptoms. Not Tested (Other): Participant suspects that they've been exposed to COVID-19, but have not shown symptoms and wonder if they have antibodies so they may return to some normalcy.
  Interventions: Device: Premier Biotech COVID-19 IgG/IgM Rapid test Cassette

INTERVENTIONS:
Device: Premier Biotech COVID-19 IgG/IgM Rapid test Cassette — Current emergency situation, there are large numbers of COVID-19 Antibody tests being made available at a record pace.
  The protocol is designed to be test agnostic. However, for this first volley, we have chosen the The COVID-19 IgG and IgM Rapid Test provided by Premier Biotech.
  We chose the Precision Bio test for 4 reasons
  1. It is available as a single use test kit in one sealed unit.
  2. It's a rapid test, with results available in 10 minutes.
  3. It has clear and easy to read instructions already included
  4. It has one of the lowest false positive rates of known tests at the moment

SUMMARY:
Radish Health and ProofPilot in coordination with Sanesco are running this study to help establish whether the Premier Biotech COVID-19 IgG/IgM Rapid Test Cassette (Whole Blood/Serum/Plasma Authorized for distribution under emergency use authorization - though not yet FDA reviewed) can be conducted effectively at home to detect COVID-19 antibodies among individuals who have tested positive, or suspect they have previous contracted from COVID-19 and recovered. The study also aims to examine how the results of those tests change social-distancing behaviors and general anxiety over 8 weeks post-test.

ELIGIBILITY:
Inclusion Criteria:

* Reside and Currently in New York City
* Does not have a blood clotting disease
* Is not abnormally queasy about taking a blood sample
* Not on any blood thinning medications
* Able to consent
* Willingness to take a blood sample
* Confirmed of highly likely past infection with COVID-19 over 14 days ago and fully recovered

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-07-29 (Estimated); Study Completion 2020-08-29 (Estimated)

PRIMARY OUTCOMES:
Does Participant Accurately Read Result | Day 0
  Comparison of participant reported self-test result vs physician review of self-test results via participant reported photograph of the test
Acceptability and Usability of Tests | Day 0
  Mesure of participant self report on ease of test administration via a custom survey assessment

SECONDARY OUTCOMES:
Social Distancing Behavior Change | Week 8
  Change in Actual vs Anticipated social distancing behavior as measured by modified PROMIS Satisfaction with Social Questionnaire.
COVID-19 Related Anxiety | Week 8
  Change in economic, personal and other anxiety triggers as measured by a modified version of the Zung Self-Rating Anxiety Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot Online App (https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Given the enormous policy and health implications, we will be making results available as soon as there are sufficient data sets to analyze. We will also provide our study design for replication in other environments and via other tests.
Supporting Information: Study Protocol, ICF
Time Frame: As soon reasonably sized data sets are available.
Access Criteria: No personally identifiable information will be provided. Those who wish to access must have a ProofPilot account. All access must be approved by study investigators.
URL: http://go.proofpilot.com